CLINICAL TRIAL: NCT05518266
Title: Ultrasound-guided Versus Surgeon Delivered Post-incisional Parasternal Block in Adult Patients Undergoing Open Cardiac Surgery: Are They the Same?
Brief Title: Sonar Guided vs Surgeon Delivered Parasternal Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Ali Ahmed, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIFPB Adults
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Parasternal Intercostal Nerve Block
Keywords: pectointercostal fascial plane block; parasternal block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-guided post-incisional PIFB (Active Comparator): Bupivacaine 0.25 % will be injected into the fascial plane between the pectoralis major muscle and external intercostal muscle or costal cartilages on each side of the sternum after skin closure under ultrasound guidance
  Interventions: Procedure: US-guided Parasternal block
- Surgeon-delivered post-incisional parasternal block (Active Comparator): Just before wiring the sternum, the surgeon will inject bupivacaine 0.25 % in 4 mL aliquots into the anterior (2nd-6th) intercostal spaces on each side about 2 cm lateral to the sternal edge with a total volume of 40 mL under direct vision.
  Interventions: Procedure: Surgeon-delivered parasternal block

INTERVENTIONS:
Procedure: US-guided Parasternal block — Bupivacaine 0.25 % will be injected into the fascial plane between the pectoralis major muscle and external intercostal muscle or costal cartilages on each side of sternum after skin closure under ultrasound guidance
  Other Names: Pectointercostal fascial plane block
  Arms: US-guided post-incisional PIFB
Procedure: Surgeon-delivered parasternal block — Just before wiring of the sternum, the surgeon will inject bupivacaine 0.25 % in 4 mL aliquots into the anterior (2nd-6th) intercostal spaces on each side about 2 cm lateral to the sternal edge with a total volume of 40 mL under direct vision.
  Arms: Surgeon-delivered post-incisional parasternal block

SUMMARY:
The objective of this study is to determine whether the use of post-incisional surgeon-delivered parasternal block is at least non-inferior in relieving postoperative pain in adult patients scheduled for cardiac surgery involving sternotomy compared with ultrasound-guided post-incisional PIFB.

DETAILED DESCRIPTION:
Patients will be randomly allocated (using a sequence of computer-generated random numbers) into one of two groups (44 patients in each); group P (ultrasound guided parasternal; PIFP block) and group S (surgeon delivered parasternal block).

1. group P (ultrasound guided parasternal; PIFP block): Bupivacaine 0.25 % will be injected into the fascial plane between the pectoralis major muscle and external intercostal muscle or costal cartilages on each side of sternum after skin closure under ultrasound guidance
2. Group S (surgeon delivered parasternal block). Just before wiring the sternum, the surgeon will inject bupivacaine 0.25 % in 4 mL aliquots into the anterior (2nd-6th) intercostal spaces on each side about 2 cm lateral to the sternal edge with a total volume of 40 mL under direct vision.

ELIGIBILITY:
Inclusion Criteria:

* Age: from 18 to 75 years.
* Rheumatic heart disease needing elective valve replacement (mitral, aortic, or double valve replacement) via median sternotomy and under CPB (cardiopulmonary bypass)
* Hemodynamic stability (no evidence of heart failure, not on vasoactive drugs, and not on mechanical ventilation).

Exclusion Criteria:

* • Previous, urgent, or emergent cardiac surgery.

  * Patients undergoing coronary artery bypass grafting (CABG)
  * local infection of the skin at the site of needle puncture,
  * Allergy to bupivacaine,
  * Coagulation disorders,
  * Clinically significant liver or kidney disease,
  * Heart failure or severe pulmonary hypertension.
  * severe renal, pulmonary, liver, or endocrine systemic disease,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative pain score | 24 hours
  Postoperative pain score will be measured after extubation at 0, 3, 6, 12, 16, 20, and 24 hours, using a visual analog scale (VAS). We are interested in the time at which postoperative pain is most severe.
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually, 10centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme.
  A score of 0 is "no pain and a score of 10 is "worst imaginable pain"

SECONDARY OUTCOMES:
Amount of rescue analgesia | 24 hours
  Amount of rescue analgesia (total dose of fentanyl) during the first 24 hours after extubation.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Result] Huang AP, Sakata RK. [Pain after sternotomy - review]. Rev Bras Anestesiol. 2016 Jul-Aug;66(4):395-401. doi: 10.1016/j.bjan.2014.09.003. Epub 2015 Mar 18. Portuguese. PMID 25796483
- [Result] Vilite B, Strike E, Rutka K, Leibuss R. Pain management in intensive care unit patients after cardiac surgery with sternotomy approach. Acta Med Litu. 2019;26(1):51-63. doi: 10.6001/actamedica.v26i1.3956. PMID 31281217